CLINICAL TRIAL: NCT03114397
Title: Long-term Effect of 20 Sessions of Transcranial Direct Current Stimulation in Patients With Disorders of Consciousness: a Double Blind Sham Controlled Clinical Trial.
Brief Title: Long-term Effect of tDCS in Patients With Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Fondazione Salvatore Maugeri, Italy (Unknown); Université Catholique de Louvain, Belgium (Unknown); Hospitales Nisa, Spain (Unknown); I.R.C.C.S. Fondazione Santa Lucia, Italy (Unknown); Schoen Clinic Bad Aibling, Germany (Unknown); Research Center of Neurology, Russia (Other Government); Therapiezentrum Burgau, Germany (Unknown); pavlov state medical university, Russia (Unknown); Azienda Unita Sanitaria Locale di Piacenza, Italy (Unknown)
Responsible Party: Principal Investigator, Aurore Thibaut, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/113b
Record Dates: First submitted 2017-03-29; First posted 2017-04-14 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Disorder of Consciousness
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal stimulation (Active Comparator): Patients will receive anodal tDCS (on the left dorsolateral prefrontal cortex) every day for 4 weeks, 5 days per week (tDCS of 2mA during 20minutes) for a total of 20 sessions.
  Interventions: Device: transcranial direct current stimulation - active
- sham stimulation (Placebo Comparator): Patients will receive sham tDCS (on the left dorsolateral prefrontal cortex) every day for 4 weeks, 5 days per week (tDCS of 2mA during 20minutes) for a total of 20 sessions.
  Interventions: Device: transcranial direct current stimulation - sham

INTERVENTIONS:
Device: transcranial direct current stimulation - active — transcranial direct current stimulation will be applied over the left dorsolateral at 2 mA for 20minutes.
  Arms: anodal stimulation
Device: transcranial direct current stimulation - sham — transcranial direct current stimulation will be applied over the left dorsolateral at 2 mA for 20minutes. The sham intervention consists of 30 seconds of stimulation at the beginning and the end of the 20minutes of intervention.
  Arms: sham stimulation

SUMMARY:
In this multicentric double-blind sham controlled study, the investigators plan to assess the effects of 20 sessions of tDCS on long-term behavioral recovery in patients with disorders of consciousness. Neurophysiological outcomes (EEG) will also be collected.

This research will 1) determine whether long-term behavioral recovery can be promoted with tDCS and 2) generate knowledge regarding the impact of tDCS on neurophysiological outcome (i.e., EEG) in severely brain injured patients. The investigators will compare the effects of active and sham tDCS on behavioral assessments and quantitative EEG in patients with severe brain injury and its potential application in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* CNS medication stable for at least a week
* Stable diagnosis (no diagnosis change based on 2 CRS-R performed within 1 week).
* Between 3 and 24 months post injury
* Structural MRI or CT-scan (to evidence focal lesions on the left DLPFC)

Exclusion Criteria:

* Craniotomies encompassing the frontal region (electrodes location)
* VPS under the stimulated area (prefrontal cortex)
* Pacemaker
* Metallic cerebral implant
* Severe medical conditions that might influence clinical diagnosis and EEG activity (e.g., severe hepatic insufficiency or renal failure, or sub-continuous or abundant epileptiform discharges on standard EEG recordings).

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R total score | 4 weeks
  Improvement of the CRS-R total score after the end of the anodal session.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liege, Liège, Belgium

REFERENCES:
- [Background] Thibaut A, Wannez S, Donneau AF, Chatelle C, Gosseries O, Bruno MA, Laureys S. Controlled clinical trial of repeated prefrontal tDCS in patients with chronic minimally conscious state. Brain Inj. 2017;31(4):466-474. doi: 10.1080/02699052.2016.1274776. Epub 2017 Mar 10. PMID 28281845
- [Background] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549